CLINICAL TRIAL: NCT00699062
Title: Effect of Montelukast on the Airway Remodeling in Asthma Patients: Physiological-radiological Correlation
Brief Title: Effect of Montelukast on the Airway Remodeling
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jinming Gao, Professor of Pulmonary Medicine, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JGao001; Merck-IISP001 (Other Grant/Funding Number: MSD pharmaceutical)
Record Dates: First submitted 2008-06-11; First posted 2008-06-17 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Asthma
Keywords: antileukotriene; small airway; airway remodeling; HRCT
MeSH Terms: conditions — Asthma; Airway Remodeling | interventions — Single Person; montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo pill (Placebo Comparator): The patients allocated into this placebo comparator arm will receive inhale corticosteroid plus long-acting bronchodilator plus placebo for 6 months.
  Interventions: Drug: placebo
- Singular pill (Experimental): The patients in this placebo comparator arm will receive inhale corticosteroid plus long-acting bronchodilator and montelukast for 6 months
  Interventions: Drug: singular

INTERVENTIONS:
Drug: singular — The participants randomized into this arm will receive singular 10mg q.n. plus combine therapy with inhaled ICS+LABA
  Other Names: montelukast
  Arms: Singular pill
Drug: placebo — The participants allocated into this arm will receive placebo 10mg,q.n plus combine therapy with inhaled ICS+LABA
  Arms: Placebo pill

SUMMARY:
The distal lung contributes to asthmatic airway remodeling which is observed from early onset of the disease. Cysteinyl leukotrienes (CysLT) play important role in the pathogenesis of airway remodeling and antileukotrienes work to exert a certain degree of anti-inflammatory effect. The cysteinyl leukotriene antagonist Montelukast has been in vivo shown to significantly inhibit ovalbumin induced airway smooth muscle hyperplasia and subepithelial fibrosis in sensitized mice. This study aims to evaluate if Montelukast could reverse airway remodeling in asthma patients by a non-invasive approach-HRCT.

DETAILED DESCRIPTION:
Accumulated data have suggested that the distal lung, which includes airways of < 2mm in diameter and lung parenchyma, contribute to asthma pathogenesis and symptoms. In addition to persisting inflammation, distal lung undergoes remodeling, as demonstrated by the reduced elastic fiber content and abnormal alveolar attachments, with the latter thought to result in a loss of elastic recoil and a reduction in FEV1.0. Furthermore, recent studies have shown that airway remodeling is observed from early onset of the disease and may, therefore, be characteristic of asthma. Amounting evidence has revealed that airway remodeling of asthmatic airways accounts for a large component of airway hyperresponsiveness (AHR) and excessive airway narrowing.

Since remodeling processes occur in parallel to, or may even be obligatory for, the establishment of persistent inflammation, the pathogenesis of airway remodeling and the implications of therapeutic interventions that are designed to diminish airway remodeling remain important areas of both research and clinic. Inhale corticosteroid (ICS) is mainstay for the treatment of asthma, however, ICS provides very little benefit for airway remodeling.

Cysteinyl leukotrienes (CysLT) play important role in the pathogenesis of airway remodeling and antileukotrienes work to exert a certain degree of anti-inflammatory effect. The cysteinyl leukotriene antagonist Montelukast, for example, has been in vivo shown to significantly inhibit ovalbumin induced airway smooth muscle hyperplasia and subepithelial fibrosis in sensitized mice. Montelukast, a systemically delivered leukotriene receptor antagonist, has been strongly recommended to treat asthma by several guidelines. Clinically, the systemically acting oral agent montelukast has been shown to improve proximal and distal lung physiology. In particular, improvements in distal lung function correlate with improvements in asthma symptoms. The in vivo experiments performed in rodent animal challenged by OVA have shown that Montelukast can reverse airway remodeling, as well as inhibit inflammation.

To determine the occurrence of airway remodeling in human being, bronchial biopsy samples obtained with a bronchoscope are subjected to histological examination. However, bronchial biopsy is invasive and causes considerable pain, while assessment of the peripheral small airways and of changes in the deep submucosal tissue and airway smooth muscle in large airways is technically difficult. This technique does not allow the longitudinal analysis of airway wall dimensions.

Noninvasive evaluation of airways by means of imaging with high-resolution computed tomography (HRCT) has therefore been tried as an alternative procedure, and was found to have the potential to evaluate airways in patients with obstructive pulmonary disease. The measurement of airway wall thickness by HRCT in patients with asthma has been demonstrated to correlate with the severity of asthma. Computed tomographic imaging of the airways by HRCT has been widely applied to investigate the alterations in the structure of the airways termed airway remodeling in patients with airway obstructive diseases (see references 1-4).

So far to our knowledge, there is no study aiming to evaluate if Montelukast could reverse airway remodeling in asthma patients by HRCT.

Our encouraging preliminary data performed in 4 patients with moderate to severe asthma according to GINA definition who received oral Montelukast for 3 months demonstrate with or without combination of ICS+LABA that there were significant improvements in airway wall thickness and air trapping evaluated by measurement of HRCT and lung function in patients with oral Montelukast as compared with those without oral Montelukast. We adopted WA% and WA/BSA to reflect the degree of airway thickness as published methods. We found that the patients who received oral montelukast for 3 months experienced improvements in airway remodeling. WA/BSA and WA% significantly decreased compared to the baseline.

The purpose of the proposal presented is to further examine, in a relatively large number of patients, that Montelukast can improve the structural changes in the large airways and air trapping by means of HRCT, and their relationship with pulmonary function in patients in moderate to severe asthma.

ELIGIBILITY:
Inclusion Criteria:

* forced expiratory volume in one second (FEV1) is at 60-80% predicted or less than 60% predicted
* clinical diagnosis of moderate-to-severe asthma.

Exclusion Criteria:

* intravenous, oral or intramuscular steroids used within 1 months
* Anti-leukotrienes, cromolyn sodium or nedocromil used within 2 months
* Theophylline or beta-adrenergic blockers used within 1 month
* Tobacco Used within the past year or cumulative smoking history > 5 pack-yrs
* Respiratory infection or an influenza vaccination Within 3 weeks
* Pregnant or lactating females
* Patient has a history of an anaphylactic allergic reaction related to administration of either a marketed or investigational drug

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To evaluate distal airway function using high-resolution CT and lung function test | 6 months
  To demonstrate that the correlation between non-invisive chest HRCT and lung function test in patients moderate-to-severe asthma

SECONDARY OUTCOMES:
Montelukast can bring additional benefit for lung function improvement in moderate to severe patients with asthma | 6 months
  To test whether montelukast can improve the distal airway function

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Gao, M.D., Ph.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

REFERENCES:
- [Background] Henderson WR Jr, Chiang GK, Tien YT, Chi EY. Reversal of allergen-induced airway remodeling by CysLT1 receptor blockade. Am J Respir Crit Care Med. 2006 Apr 1;173(7):718-28. doi: 10.1164/rccm.200501-088OC. Epub 2005 Dec 30. PMID 16387808
- [Background] Gono H, Fujimoto K, Kawakami S, Kubo K. Evaluation of airway wall thickness and air trapping by HRCT in asymptomatic asthma. Eur Respir J. 2003 Dec;22(6):965-71. doi: 10.1183/09031936.03.00085302. PMID 14680087
- [Background] Mitsunobu F, Ashida K, Hosaki Y, Tsugeno H, Okamoto M, Nishida N, Nagata T, Takata S, Tanizaki Y. Decreased computed tomographic lung density during exacerbation of asthma. Eur Respir J. 2003 Jul;22(1):106-12. doi: 10.1183/09031936.03.00081702. PMID 12882459
- [Background] Zeidler MR, Kleerup EC, Goldin JG, Kim HJ, Truong DA, Simmons MD, Sayre JW, Liu W, Elashoff R, Tashkin DP. Montelukast improves regional air-trapping due to small airways obstruction in asthma. Eur Respir J. 2006 Feb;27(2):307-15. doi: 10.1183/09031936.06.00005605. PMID 16452585
- [Background] King GG, Muller NL, Pare PD. Evaluation of airways in obstructive pulmonary disease using high-resolution computed tomography. Am J Respir Crit Care Med. 1999 Mar;159(3):992-1004. doi: 10.1164/ajrccm.159.3.9805064. No abstract available. PMID 10051284
- [Derived] Gao JM, Cai F, Peng M, Ma Y, Wang B. Montelukast improves air trapping, not airway remodeling, in patients with moderate-to-severe asthma: a pilot study. Chin Med J (Engl). 2013 Jun;126(12):2229-34. PMID 23786930
- See also: this website provides the updated information on the this study — http://www.ncbi.nlm.nih.gov